CLINICAL TRIAL: NCT04325074
Title: Mental Practice and Manipulative Skills Training in Multiple Sclerosis: a Pilot Study
Brief Title: Mental Practice and Manipulative Skills Training in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cristina García-Bravo (Other)
Responsible Party: Sponsor-Investigator, Cristina García-Bravo, Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 220720153515
Record Dates: First submitted 2020-03-18; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mental practice (Experimental): The final sample therefore comprised of 35 participants (n=35), who were divided into three treatment groups. The sample of mental practice group was n=12.
  Interventions: Other: Mental practice
- Mental practice + skill training (Experimental): The final sample therefore comprised of 35 participants (n=35), who were divided into three treatment groups. The sample of mental practice + skills training group was n=13.
  Interventions: Other: Mental practice + skill training
- Control group (Active Comparator): The final sample therefore comprised of 35 participants (n=35), who were divided into three treatment groups. The sample of control group was n=10.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Mental practice — During each of the 12 treatment sessions, the patient was asked to select two tasks from a list of MP activities, graded by level. Once the task was selected, patients received the specific visual or audio instructions and subsequently performed the task. The recording was viewed three times and the audio instructions were repeated two times. To listen to the audio instructions, the participants were requested to close their eyes in order to aid concentration. After listening to the recordings, the patient was asked to perform the task once again, practicing what had been learnt. After the process was completed, the participant completed a questionnaire and scored each task.
  Arms: Mental practice
Other: Mental practice + skill training — In this option, six sessions of MP were alternated with six sessions of skills training (ST). The MP protocol was the same as in group A: selecting, performing, visualizing, listening to and scoring the selected tasks. The activities performed in the skills training were based on the Kamm et al. (2015) protocol and bimanual tasks. After the performance of each task, the patients were allowed to rest for 1 or 2 minutes to avoid the appearance of fatigue.
  Arms: Mental practice + skill training
Other: Control group — The control group only received their usual physical therapy and occupational therapy treatments provided by their association. The treatment mainly consisted of the application of the Bobath concept and the Vojta method, dry needling, myofascial induction therapy, passive mobilizations, training of gross and fine motor coordination of the upper limbs, resistance training and static and dynamic balance training.
  Arms: Control group

SUMMARY:
Introduction: Multiple sclerosis (MS) is a demyelinating disease of the central nervous system which produces both motor and cognitive dysfunctions. MS causes a decline in the performance of activities of daily living (ADL) due to impairments affecting limb function.

Aim: This pilot study sought to determine whether the use of mental practice (MP) or the combined use of MP and the training of manipulative skills would improve the manipulation motor skills and treatment satisfaction among people with MS.

Methods: The study participants were people with MS. Blinded evaluators performed three assessments for each patient (pre-treatment, post-treatment and at a three month follow up). The patients were divided into three groups with alternate allocation: (A) Mental practice, (B) Mental practice + skills training and (C) Control group.

Keywords: activities of daily living; manual dexterity; mental practice, motor image; multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with MS of the RRMS and SPMS subtypes, without the presence of flare-ups during the past three months and aged between 25 and 60 years;
* an Expanded Disability Status Scale (EDSS) score of ≤7,
* not presenting depressive symptoms (measured using the Beck Depression Inventory, BDI),
* not presenting cognitive decline, measured using the Montreal Cognitive Assessment (MoCA) or Minimental Status Examination.
* In addition, they had to be regularly attending physical therapy and/or occupational therapy rehabilitation treatments.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Nine Hole Peg Test (NHPT). Pre-treatment | Pre-treatment assessments were performed with each patient.
  The higher scores mean a worse outcome.
Box and Block Test (BBT). Pre-treatment | Pre-treatment assessments were performed with each patient.
  The higher scores mean a better outcome.
The ABILHAND questionnaire. Pre-treatment | Pre-treatment assessments were performed with each patient.
  The higher scores mean a better outcome.
The Canadian Occupational Performance Measure (COPM). Pre-treatment | Pre-treatment assessments were performed with each patient.
  The higher scores mean a better outcome.

SECONDARY OUTCOMES:
Nine Hole Peg Test (NHPT). Post-treatment | Immediately after treatment assessments were performed with each patient.
  The higher scores mean a worse outcome.
Box and Block Test (BBT). Post-treatment | Immediately after treatment assessments were performed with each patient.
  The higher scores mean a better outcome.
The ABILHAND questionnaire. Post-treatment | Immediately after treatment assessments were performed with each patient.
  The higher scores mean a better outcome.
The Canadian Occupational Performance Measure (COPM). Post-treatment | Immediately after treatment assessments were performed with each patient.
  The higher scores mean a better outcome.

OTHER OUTCOMES:
Nine Hole Peg Test (NHPT). Three-month follow-up | Three-month follow-up assessments were performed with each patient.
  The higher scores mean a worse outcome.
Box and Block Test (BBT). Three-month follow-up | Three-month follow-up assessments were performed with each patient.
  The higher scores mean a better outcome.
The ABILHAND questionnaire. Three-month follow-up | Three-month follow-up assessments were performed with each patient.
  The higher scores mean a better outcome.
The Canadian Occupational Performance Measure (COPM). Three-month follow-up | Three-month follow-up assessments were performed with each patient.
  The higher scores mean a better outcome.

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be sent by email.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At present
Access Criteria: cristina.bravo@urjc.es